CLINICAL TRIAL: NCT00840463
Title: Safety and Efficacy Trial Using Ambrisentan for Pulmonary Hypertension Associated With Congestive Heart Failure With Preserved Left Ventricular Ejection Fraction
Brief Title: Safety and Efficacy Trial to Treat Diastolic Heart Failure Using Ambrisentan
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrolment
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IN-US-300-0126
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Hypertension; Heart Failure With Preserved Ejection Fraction
Keywords: Pulmonary Hypertension; Diastolic Heart Failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure, Diastolic | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Ambrisentan
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Subjects will be initiated at 2.5 mg per day and increased to 5mg daily in 2 weeks and then 10mg daily if clinically tolerated (edema is controlled and symptoms are stable).
  Other Names: Letairis
  Arms: 1
Other: Placebo — Sugar pill
  Other Names: The placebo will look identical to the Ambrisentan tablets
  Arms: 2

SUMMARY:
This is a randomized study of ambrisentan that will last 16 weeks. The study will include patients with diastolic heart failure and pulmonary hypertension. Patients will be randomized (1:1) to ambrisentan or placebo. The ambrisentan or matching placebo will be started at 2.5 mg by mouth daily and increased to 5mg and then 10mg daily, if tolerated. Patients will be seen at least monthly for 16 weeks. Adverse reactions will be reviewed and the required monthly laboratory tests (liver function testing and pregnancy testing, if applicable), will be performed. Patients will also complete an exercise test (six minute walk distance) and a quality of life survey at the baseline, week 4 and week 16 visit. An echocardiogram and a right heart catheterization and left ventricular end diastolic pressure measurement will be performed at the 16 week visit. The primary end-point is safety, and secondary end-points include the catheterization results, echocardiogram results, the walk distance and the quality of life survey. The expected completion of the study is 18 months from initiation. Ambrisentan is an FDA approved drug for PAH, but not for CHF.

DETAILED DESCRIPTION:
Hypothesis: patients with pulmonary hypertension secondary to diastolic congestive heart failure (CHF) treated with ambrisentan for 16 weeks will have improved hemodynamics, increased exercise capacity and improved functional class with an acceptable safety profile, compared with placebo treated patients.

Objectives: to evaluate the safety and efficacy of ambrisentan treatment in patients with pulmonary hypertension due to diastolic CHF. Efficacy will be assessed by improvement in hemodynamics (PVR(Pulmonary Vascular Resistance): primary efficacy endpoint), six minute walk distance (6MWD), World Health Organization (WHO) functional class and quality of life after 16 weeks of treatment with ambrisentan. Safety of ambrisentan will be compared to placebo.

Concomitant Medication: Treatment with standard medications for CHF including diuretics and optimal blood pressure control with antihypertensive medications will be allowed throughout the study period. Diuretics adjustment will also be allowed and encouraged based on the planned diuretic management protocol. Approved medications for CHF in general are allowed as well, though it should be noted that there are no medications shown to have benefit in diastolic CHF. Patients may not be on an endothelin antagonist or sildenafil.

ELIGIBILITY:
Inclusion Criteria:

1. Catheterization

   1. Elevated pulmonary arterial pressure (PA mean >25mmHg)
   2. Elevated pulmonary vascular resistance (>240 dynes.cm.sec-5) or transpulmonary gradient (>12 mmHg)
   3. Elevated LVEDP (>15mmHg, but ≤23 mmHg)
2. Evidence of left ventricular diastolic dysfunction: LA>4.0, LVH or diastolic dysfunction by mitral filling pattern
3. Echocardiogram: Normal or mildly reduced LV ejection fraction (greater than or equal to 40%)
4. Symptomatic chronic HF (WHO functional class II-IV)
5. Baseline walk distance 100 to 400 meters
6. Age 18 - 80 (increased from 70)

Maximal treatment of diastolic dysfunction as noted by the treating physicians with no change in medical therapy for one month prior to entry

Exclusion Criteria:

1. Use of endothelin receptor antagonist, prostacyclin or PDE-5 inhibitor within 4 weeks of enrollment
2. Exercise capacity limited by other illness (other lung disease, arthritis, mobility limitations)
3. Uncontrolled systemic hypertension
4. Uncontrolled atrial fibrillation
5. Severe valvular disease
6. Pregnant females- females of child bearing potential will need to use contraceptive agent barrier given the teratogenicity associated with ERA's
7. Uncontrolled OSA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Chin, MD, Principal Investigator — University of Texas Southwestern Medical Center; Fernando Torres, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through the UTSW clinics. Recruitment difficulties arose and the study was halted due to poor recruitment
Period: Overall Study
Arm/Group | Ambrisentan | Placebo
Started | 3 | 1
Completed | 2 | 1
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan | Placebo | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [57 to 66] | 50 [50 to 50] | 59.5 [52 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance (Wood Units)
Description: The primary efficacy outcome will be Pulmonary Vascular Resistance.PVR will be calculated as [(PA mean - wedge) / Cardiac Output]
Time Frame: Baseline and Four months
Measure: Mean (Full Range); unit: wood units
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 2 | 1
wood units | -0.75 [-0.77 to -0.72] | 2.81 [2.81 to 2.81]

2. Primary Outcome: Safety Assessment-Number of Subjects Who Are Free and Those Who Developed Clinically Significant Adverse Events (CSAEs)
Description: Freedom from clinically significant adverse events will be measure by determining the number free from CSAEs and those who developed CSAEs
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 3 | 1
Participants
  Free from clinically significant AE | 2 | 1
  Developed clinically significant AE | 1 | 0

3. Secondary Outcome: Change in 6 Minute Walk Distance
Description: subjects complete the 6 minute walk test to determine how far (in meters) they are able to walk in 6 minutes.
Time Frame: Baseline and Four months
Measure: Mean (Full Range); unit: meters
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 2 | 1
meters | -22 [-93 to 48] | 53 [53 to 53]

4. Secondary Outcome: Change in Functional Class
Description: Change in functional class from baseline to month 4. This is graded from WHO FC I to FC IV. Assessment will be completed by an investigator on the study at every visit.
Time Frame: basline and 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 3 | 1
Participants
  Improved | 0 | 0
  Stable | 3 | 1
  Worsened | 0 | 0

5. Secondary Outcome: Change in Short Form-36 Physical Functioning
Description: Change between baseline and follow-up in the physical functioning items of the SF-36 questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health
Time Frame: baseline 4 months
Population: note that there was no change in the SF-36 score (baseline to month 4) for the placebo arm hence the mean is not meaningful
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 2 | 1
score on a scale | 12.5 [-10 to 35] | 0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | Ambrisentan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (N=3) | Placebo (N=1)
Admission for heart failure (Cardiac disorders) | 1 (1) | 0 (0) — Developed dyspnea and 15 pound weight gain requiring admission for diuresis during week 8 of the study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (N=3) | Placebo (N=1)
Edema (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain or tightness (Cardiac disorders) | 2 (2) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No